CLINICAL TRIAL: NCT01113528
Title: The Effect of Host Response Modulation Therapy (Omega 3 Plus Low-dose Aspirin) as an Adjunctive Treatment of Chronic Periodontitis (Clinical and Biochemical Study)
Brief Title: Omega-3 and Aspirin in Periodontal Regeneration
Acronym: PR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Amr Moustafa Elkhouli, Lecturer, O6U
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHDA-1962; October 6 U 196222 (Other: October 6 University)
Record Dates: First submitted 2010-04-23; First posted 2010-04-30 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Periodontal Disease
Keywords: Bone allograft; IL-1; IL-10; periodontal regeneration; omega-3; aspirin
MeSH Terms: conditions — Periodontal Diseases | interventions — Aspirin; Fish Oils; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regenerative therapy (Experimental)
  Interventions: Other: Regenerative therapy (omega 3 PUFA plus low dose aspirin)
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Other: Regenerative therapy (omega 3 PUFA plus low dose aspirin) — Comparison between regenerative bone graft alone and bone graft + Omega-3 and low dose aspirin
  Other Names: Omega; Fish oil; ASA; low dose aspirin; DFDBA
  Arms: Regenerative therapy
Drug: Sugar pill — 3 times daily
  Other Names: Gelatinous capsules
  Arms: Sugar pill

SUMMARY:
To evaluate the efficacy of systemic administration of omega 3 PUFA plus low dose aspirin as an adjunctive therapy to regenerative modality of grade II furcation defects in periodontitis patients.

DETAILED DESCRIPTION:
In this study, we tested the hypothesis that the administration of omega 3 PUFA plus low dose aspirin would augment the results following regenerative therapy of furcation defects in chronic periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* suffering moderate to sever chronic periodontitis and displaying at least a single grade II furcation defect according to Glickman's classification 1953, determined by both clinical and radiographic examinations;
* free from systemic diseases known to influence the periodontal condition and not receiving any medication known to affect the periodontal status;
* have not receive any periodontal therapy for a minimum of 6 months prior to the study.

Exclusion Criteria:

* Known hypersensitivity or allergy to one of the used medications
* Pregnancy or lactation
* Heavy smoking (more than 10cigarretes/day)
* History of alcohol abuse
* Participation in other clinical trials

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Cytokine levels | six months
  Interleukin-1 beta Interleukin-10

SECONDARY OUTCOMES:
Gingival inflammation | six months
  plaque index Gingival index Gingival bleeding index
Healing after regenerative therapy | six months
  Probing pocket depth Clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Amr M. Elkhouli, ph.D, Principal Investigator — October 6 University
Locations (1):
- October 6 University, Cairo, Overnorate of 6 October, Egypt